CLINICAL TRIAL: NCT06576141
Title: The Effect of Kaleidoscope and Virtual Reality Glasses on Pain and Anxiety Levels in Venous Blood Collection in Children Aged 9-12
Brief Title: Kaleidoscope Virtual Reality Glasses Pain and Anxiety Levels in Venous Blood Collection Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, Tuğba OLUÇ, Research Assistant, Erzincan Binali Yildirim Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EBYU-SBF-TO-01
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Child, Only
Keywords: PAİN; Kaleidoscope; Venous Blood Collection; Anxiety; Virtual Reality Glasses; Children
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: There are three groups. Kaleidoscope ,Virtual Reality Glasses and control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will be done via random.org.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kaleidoscope group (Active Comparator): The kaleidoscope will be used 5 minutes before the blood collection procedure, as the child who will be included in the kaleidoscope group sits in the patient chair. The nurse will start preparing the child for the blood collection procedure at that time.
  Interventions: Other: Kaleidoscope
- virtual reality glasses (Active Comparator): The child to be included in the virtual reality group will be seated in the patient chair and the virtual reality will be used 5 minutes before the blood collection procedure. The nurse will start preparing the child for the blood collection procedure at that time.
  Interventions: Other: Virtual Reality
- control group (Other): Children in the control group will not undergo any interventional procedures. Blood collection will be arranged to be taken from the antecubital region by the same nurse via a vacutainer.
  Interventions: Other: control

INTERVENTIONS:
Other: Kaleidoscope — The participation of patients in this group in the study will take approximately 15-20 minutes.
  Arms: Kaleidoscope group
Other: Virtual Reality — The participation of patients in this group in the study will take approximately 15-20 minutes.
  Arms: virtual reality glasses
Other: control — The participation of patients in this group in the study will take approximately 5-10 minutes.
  Arms: control group

SUMMARY:
The aim of our research is to investigate the effects of distracting children's attention with a kaleidoscope and virtual reality glasses during venous blood collection on perceived pain and anxiety levels.

DETAILED DESCRIPTION:
After obtaining the necessary institutional permissions, parents and children who come to the blood collection room will be informed about the research through the "Informed Consent Form". The research data will be collected by the researcher using a face-to-face interview technique. Before the blood collection procedure, the children and their families who will be included in the kaleidoscope group, virtual reality group and control group will be informed about the research. The kaleidoscope will be used 5 minutes before the blood collection procedure as the child who will be included in the kaleidoscope group sits in the patient chair. The nurse will start preparing the child for the blood collection procedure at that time. The nurse will apply a tourniquet and determine the vein from the antecubital region to be taken from. The blood collection procedure will be taken from the antecubital region by the same nurse in one go using a vakuteynir (vacuum blood collection tube) and blood coming to the Vakuteynir within 5 seconds will indicate that the procedure was successful. This procedure will take approximately 2-3 minutes and the children will watch the kaleidoscope throughout the procedure. After the procedure is completed, the children will be taken out of the blood collection room and taken to the waiting area and the children will be asked to determine the level of pain they felt during the procedure. The child will assess how much fear the child experienced during the blood collection procedure and the level of anxiety.

The child who will be taken into the virtual reality group will be seated in the patient chair and virtual reality will be used 5 minutes before the blood collection procedure. The nurse will start preparing the child for the blood collection procedure at that time. The nurse will perform the tourniquet application and the determination of the vein from the antecubital region from which the blood will be taken. The blood collection procedure will be performed by the same nurse in one go from the antecubital region using a vakutainer (vacuum blood collection tube) and blood coming into the vakutainer within 5 seconds will indicate that the procedure was successful. This procedure will take approximately 2-3 minutes and the children will be shown virtual reality throughout the procedure. After the procedure is completed, the children will be taken out of the blood collection room and taken to the waiting area and the children will be asked to determine the level of pain they felt during the procedure. The child will assess how much fear the child experienced during the blood collection procedure and the level of anxiety they experienced. Children in the control group will not undergo any interventional procedures. Blood collection will be arranged to be taken from the antecubital region by the same nurse via a vacutainer. After the procedure is completed, children will be taken out of the blood collection room and taken to the waiting area. After being allowed to rest for 1-2 minutes, a questionnaire will be administered to the children. The child will evaluate how much fear the child has during the blood collection procedure and what their anxiety is. Children in the control group will not undergo any interventional procedures.

ELIGIBILITY:
Inclusion Criteria:

The child must be between the ages of 9-12, The child and parents must agree to participate in the research, The child must be able to communicate and be open to communication, The child must not have any hearing, speech or vision disorders

Exclusion Criteria:

The child is not within the age range specified above The child and parents do not agree to participate in the research. The child has a communication problem The child has a hearing, speech or vision disorder.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Facial Expression Rating Scale (WB-FRS) | 1 year
  measuring fear
State-Trait Anxiety Inventory for Children | 1 year
  measuring anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- To Sakarya University Training and Research Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No